CLINICAL TRIAL: NCT03058263
Title: The Effectiveness of Neostigmine on the Recovery of Rocuronium-Induced Neuromuscular Blockade: A Comparison Between Partial Dose and TOF Ratio-Based Adjustment Dose
Brief Title: Effect of Neostigmine on the Recovery of Rocuronium: A Comparison Between Partial and TOF Ratio-Based Dose
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Arif H. M. Marsaban, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes011
Record Dates: First submitted 2017-02-12; First posted 2017-02-20 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Muscle Relaxant; General Anesthesia
MeSH Terms: conditions — Muscle Hypotonia | interventions — Neostigmine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- partial dose of neostigmine (Experimental): Those who received partial dose of neostigmine as rocuronium reversal
  Interventions: Drug: Dose of Neostigmine
- TOF ratio-based dose of neostigmine (Experimental): Those who received TOF ratio-based dose of neostigmine as rocuronium reversal
  Interventions: Drug: Dose of Neostigmine

INTERVENTIONS:
Drug: Dose of Neostigmine — Subjects were given partial dose of neostigmine as rocuronium reversal after the surgery had finished; subjects were given TOF ratio-based dose of neostigmine after the surgery had finished
  Other Names: prostigmin

SUMMARY:
This study aimed to evaluate the effect of Neostigmine partial dose towards neuromuscular blockade of rocuronium

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine University of Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study and randomized into two groups. Intravenous (IV) cannula with Ringer Lactate fluid, non-invasive blood pressure monitor, electrocardiogram (ECG) and pulse-oxymetry were set on the subjects in the operation room. After preoxygenation was given with 100% oxygen, general anesthesia induction was done with midazolam 0.01-0.02 mg/kg, fentanyl 3 mcg/kg, propofol 1-2 mg/kg, and rocuronium 0.6 mg/kg. Following induction, endotracheal intubation or laryngeal mask insertion was performed. Maintenance was done by sevoflurane 1.2 vol%, and fentanyl 1.2 mcg/kg. After the surgery had finished, fentanyl drip was stopped. Subjects were then observed until spontaneous breaths occured adequately (tidal volume ≥ 5 ml/kg) before train of four (TOF) ratio was evaluated using acceleromyography (AMG). Before reversal (neostigmine) was given, anesthetic gas was stopped and duration of operation as well as post-operative TOF ratio was recorded. The time since reversal was given then recorded. Group A received neostigmine partial dose (0.02 mg) in combination with atropine 0.4 mg for every milligram of neostigmine. Group B received TOF ratio-based dose of neostigmine in combination with atropine 0.4 mg for every milligram of neostigmine. After administration of neostigmine, TOF ratio was measured every 5 minutes until TOF ratio of ≥ 90% was achieved, and finally definitive airway could be removed. For Group A, another partial dose of neostigmine was given after 10 minutes from the first reversal dose if the TOF ratio of ≥90% had not been reached. For Group B, another TOF ratio-based dose of neostigmine was given after 10 minutes from the first reversal dose if the TOF ratio of ≥90% had not been reached. Subjects were then transported to recovery room. Data was analyzed using Statistical Package for the Social Sciences (SPSS), for numerical data using unpaired T-test or Mann-Whitney-U test, for categorical data using Chi-square test or Fischer Exact's Test. Data normality was tested by Kolmogorov-Smirnov test. Significant value is p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-60 years old
* American Society of Anesthesiologists (ASA) physical status I-II who were planned to undergo any elective surgery at operating room in general anesthesia
* subjects had been explained about the study, and agreed to enroll and have signed the informed consent form

Exclusion Criteria:

* BMI ≥ 30
* had any severe kidney or liver disease
* had neuromuscular disease or asthma

Drop out Criteria:

* Duration of operation less than one hour or more than 2 hours
* during surgery received maintenance dose of neuromuscular block
* intraoperative cardiac arrest was occurred

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
TOF ratio with partial dose of neostigmine | Day 1
  Train-of-Four ratio obtained from post-operative acceleromyography after the first partial dose of neostigmine had been administrated until definitive airway device can be removed
TOF ratio with TOF ratio-based dose of neostigmine | Day 1
TOF ratio between partial dose of neostigmine and TOF ratio-based dose of neostigmine | Day 1
time needed to reach TOF ratio ≥ 90% in group with partial dose of neostigmine | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Arif HM Marsaban, Consultant, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maybauer DM, Geldner G, Blobner M, Puhringer F, Hofmockel R, Rex C, Wulf HF, Eberhart L, Arndt C, Eikermann M. Incidence and duration of residual paralysis at the end of surgery after multiple administrations of cisatracurium and rocuronium. Anaesthesia. 2007 Jan;62(1):12-7. doi: 10.1111/j.1365-2044.2006.04862.x. PMID 17156221
- [Background] Murphy GS, Brull SJ. Residual neuromuscular block: lessons unlearned. Part I: definitions, incidence, and adverse physiologic effects of residual neuromuscular block. Anesth Analg. 2010 Jul;111(1):120-8. doi: 10.1213/ANE.0b013e3181da832d. Epub 2010 May 4. PMID 20442260
- [Background] Thilen SR, Hansen BE, Ramaiah R, Kent CD, Treggiari MM, Bhananker SM. Intraoperative neuromuscular monitoring site and residual paralysis. Anesthesiology. 2012 Nov;117(5):964-72. doi: 10.1097/ALN.0b013e31826f8fdd. PMID 23001053
- [Background] Donati F. Residual paralysis: a real problem or did we invent a new disease? Can J Anaesth. 2013 Jul;60(7):714-29. doi: 10.1007/s12630-013-9932-8. Epub 2013 Apr 27. PMID 23625545
- [Background] Debaene B, Plaud B, Dilly MP, Donati F. Residual paralysis in the PACU after a single intubating dose of nondepolarizing muscle relaxant with an intermediate duration of action. Anesthesiology. 2003 May;98(5):1042-8. doi: 10.1097/00000542-200305000-00004. PMID 12717123
- [Background] Naguib M, Kopman AF, Ensor JE. Neuromuscular monitoring and postoperative residual curarisation: a meta-analysis. Br J Anaesth. 2007 Mar;98(3):302-16. doi: 10.1093/bja/ael386. PMID 17307778
- [Background] Song IA, Seo KS, Oh AY, No HJ, Hwang JW, Jeon YT, Park SH, Do SH. Timing of reversal with respect to three nerve stimulator end-points from cisatracurium-induced neuromuscular block. Anaesthesia. 2015 Jul;70(7):797-802. doi: 10.1111/anae.13044. Epub 2015 Feb 27. PMID 26580249
- [Background] Sundman E, Witt H, Olsson R, Ekberg O, Kuylenstierna R, Eriksson LI. The incidence and mechanisms of pharyngeal and upper esophageal dysfunction in partially paralyzed humans: pharyngeal videoradiography and simultaneous manometry after atracurium. Anesthesiology. 2000 Apr;92(4):977-84. doi: 10.1097/00000542-200004000-00014. PMID 10754616
- [Background] Viby-Mogensen J. Postoperative residual curarization and evidence-based anaesthesia. Br J Anaesth. 2000 Mar;84(3):301-3. doi: 10.1093/oxfordjournals.bja.a013428. No abstract available. PMID 10793585
- [Background] Brull SJ, Murphy GS. Residual neuromuscular block: lessons unlearned. Part II: methods to reduce the risk of residual weakness. Anesth Analg. 2010 Jul;111(1):129-40. doi: 10.1213/ANE.0b013e3181da8312. Epub 2010 May 4. PMID 20442261
- [Background] American Society of Anesthesiologists Task Force on Postanesthetic Care. Practice guidelines for postanesthetic care: a report by the American Society of Anesthesiologists Task Force on Postanesthetic Care. Anesthesiology. 2002 Mar;96(3):742-52. doi: 10.1097/00000542-200203000-00033. No abstract available. PMID 11873052
- [Background] Naguib M, Kopman AF, Lien CA, Hunter JM, Lopez A, Brull SJ. A survey of current management of neuromuscular block in the United States and Europe. Anesth Analg. 2010 Jul;111(1):110-9. doi: 10.1213/ANE.0b013e3181c07428. Epub 2009 Nov 12. PMID 19910616
- [Background] Naguib M, Samarkandi AH, Bakhamees HS, Magboul MA, el-Bakry AK. Histamine-release haemodynamic changes produced by rocuronium, vecuronium, mivacurium, atracurium and tubocurarine. Br J Anaesth. 1995 Nov;75(5):588-92. doi: 10.1093/bja/75.5.588. PMID 7577286
- [Background] Whalley DG, Maurer WG, Knapik AL, Estafanous FG. Comparison of neuromuscular effects, efficacy and safety of rocuronium and atracurium in ambulatory anaesthesia. Can J Anaesth. 1998 Oct;45(10):954-9. doi: 10.1007/BF03012303. PMID 9836032
- [Background] Grayling M, Sweeney BP. Recovery from neuromuscular blockade: a survey of practice. Anaesthesia. 2007 Aug;62(8):806-9. doi: 10.1111/j.1365-2044.2007.05101.x. PMID 17635429
- [Background] Kopman AF. Managing neuromuscular block: where are the guidelines? Anesth Analg. 2010 Jul;111(1):9-10. doi: 10.1213/ANE.0b013e3181cdb0a5. No abstract available. PMID 20576960
- See also: Van Pelt M, Chitilian HV, Eikerman M. Multi-faceted initiative designed to improve safety of neuromuscular blockade. APSF. 2016; 30: 45-76 — http://www.apsf.org/newsletters/pdf/Feb2016final_lores.pdf